CLINICAL TRIAL: NCT06129786
Title: Overcoming Therapy Resistance in ER+ Breast Cancer Patients: a Translational Project (OVERTuRE)
Acronym: OVERTuRE
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-10
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients presenting with a de novo diagnosis of luminal-like advanced breast cancer (ABC) or with disease recurrence after >12 months from the end of adjuvant ET, are generally candidate to a first line therapy with an aromatase inhibitor in association with a CDK4/6i. Disease recurrence in <12 months from the end of adjuvant ET defines the disease as "endocrine resistant" and identifies patients that should receive a first line therapy with the selective estrogen receptor degrader (SERD) Fulvestrant in association with the CDK4/6i Ribociclib, according to the results of the MONALEESA-3 trial.

A significant percentage of ABC patients develops a primary resistance with disease progression within the first 6 months from the beginning of the treatment. Furthermore, another relevant percentage of patients initially responding to the therapy, will later develop a secondary resistance, thus progressing after a median of 2 years from the beginning of the treatment. Thereby, it is crucial to identify biomarkers that could be predictive of a response or a resistance to ET and/or CDK4/6i, to provide the best therapeutic strategy, tailored upon both clinico-pathological and molecular characteristics.

Numerous pathways associated with resistance to CDK4/6i have been investigated by means of liquid biopsy analysis. The aim of this study is to identify potential biomarkers predictive of a clinical benefit in patients receiving a first line therapy with AI/fulvestrant (+/- LH-RH analogue) in association with a CDK4/6i for luminal-like advanced breast cancer.

DETAILED DESCRIPTION:
Patients presenting with a de novo diagnosis of luminal-like advanced breast cancer (ABC) or with disease recurrence after >12 months from the end of adjuvant ET, are generally candidate to a first line therapy with an aromatase inhibitor (+/- LH-RH analogue depending from the menopausal status) in association with a CDK4/6i. Disease recurrence in <12 months from the end of adjuvant ET defines the disease as "endocrine resistant" and identifies patients that should receive a first line therapy with the selective estrogen receptor degrader (SERD) Fulvestrant in association with the CDK4/6i Ribociclib, according to the results of the MONALEESA-3 trial.

The choice of the endocrine backbone and of the CDK4/6i is mostly influenced by the patient's clinical characteristics and by disease factors.

However, a significant percentage of ABC patients develops a primary resistance with disease progression within the first 6 months from the beginning of the treatment. Furthermore, another relevant percentage of patients initially responding to the therapy, will later develop a secondary resistance, thus progressing after a median of 2 years from the beginning of the treatment. Thereby, it is crucial to identify biomarkers that could be predictive of a response or a resistance to ET and/or CDK4/6i, to provide the best therapeutic strategy, tailored upon both clinico-pathological and molecular characteristics.

Numerous pathways associated with resistance to CDK4/6i have been investigated by means of liquid biopsy analysis. The aim of this study is to identify potential biomarkers predictive of a clinical benefit in patients receiving a first line therapy with AI/fulvestrant (+/- LH-RH analogue) in association with a CDK4/6i for luminal-like advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of adenocarcinoma of the breast with evidence of metastatic disease.
* ER positive tumor ≥ 1%
* HER2 negative breast cancer by FISH or IHC (IHC 0,1+, 2+ and/or FISH HER2: CEP17 ratio < 2.0)
* Females, 18 years of age or older
* Candidate to first-line endocrine therapy (LH-RH analogue for pre-menopausal women is allowed)
* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Diagnosis of any secondary malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* Prior endocrine therapy for metastatic disease
* Prior chemotherapy for metastatic disease
* Patients unwilling to or unable to comply with the protocol.
* Known CNS metastases

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with hormone receptor-positive ABC, considered eligible for endocrine therapy as first line endocrine treatment
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
To identify potential biomarkers predictive of a clinical benefit in patients receiving a first line therapy with AI/fulvestrant (+/- LH-RH analogue) in association with a CDK4/6i for luminal-like ABC. | up to 3 years
  Mean difference in mean VAF in most frequently mutated gene found at baseline, with respect to first evaluation after 15 days between responders (CR-PR-SD, Complete Response - Partial Response - Stable Disease) and non-responders (PD, Progressive Disease)
To identify potential biomarkers predictive of a clinical benefit in patients receiving a first line therapy with AI/fulvestrant (+/- LH-RH analogue) in association with a CDK4/6i for luminal-like ABC. | up to 3 years
  Mean difference in mean VAF in most frequently mutated gene found at baseline, with respect to 6 months evaluation between responders (CR-PR-SD, Complete Response - Partial Response - Stable Disease) and non-responders (PD, Progressive Disease)

SECONDARY OUTCOMES:
To explore the impact of ctDNA-based biomarkers in terms of treatment resistance | from first biomarker assessment until objective PD or end of follow-up, up to 3 years
  Differences in time-to-progression (TTP) probability between patients with or without selected ctDNA-based biomarkers. TTP will be defined as the time from first biomarker assessment until objective PD or end of follow-up, whichever comes first.
To explore the impact of ctDNA-based biomarkers in terms of survival | from beginning of the therapy until objective PD, death or end of follow-up, up to 3 years
  Differences in progression-free survival (PFS) between patients with or without selected ctDNA-based biomarkers. PFS will be defined as time from beginning of the therapy until objective PD, death or end of follow-up, whichever comes first.
To explore the impact of ctDNA-based biomarkers in terms of survival | from beginning of the therapy until death from any cause or end of follow-up, up to 3 years
  Differences in Overall survival (OS) between patients with or without selected ctDNA-based biomarkers. OS will be defined as time from beginning of the therapy until death from any cause or end of follow-up, whichever comes first.
Mean difference in mean VAF in most frequently mutated gene found at baseline, between baseline and progression in non-responders (PD, Progressive Disease) | up to 3 years
  Mean difference in mean VAF in most frequently mutated gene found at baseline, between baseline and progression in non-responders (PD, Progressive Disease)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Puglisi, MD,PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Barbara Belletti, PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (2):
- Italy (2):
  - Centro di Riferimento Oncologico (CRO) di aviano-IRCCS, Aviano, Pordenone
  - Azienda Sanitaria Universitaria del Friuli Centrale(ASUFC), Udine